CLINICAL TRIAL: NCT02245087
Title: Eliminate Coronary Artery Disease
Acronym: ECAD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Michael Farkouh, Chair of the Peter Munk Centre of Excellence in Multinational Clinical Trials, Peter Munk Cardiac Centre, UHN, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ECAD001
Record Dates: First submitted 2014-09-11; First posted 2014-09-19 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
Keywords: atorvastatin; coronary artery disease; myocardial infarction; stroke; revascularization
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Stroke | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Experimental): Atorvastatin(Lipitor) in addition to the usual guideline based care
  Interventions: Drug: Atorvastatin
- Guideline based care (No Intervention): Current guidelines for lipid-management in healthy middle aged men and women only.

INTERVENTIONS:
Drug: Atorvastatin — 20 mg of atorvastatin daily
  Other Names: Lipitor
  Arms: Atorvastatin

SUMMARY:
The purpose of this study is to determine whether pharmacologic lowering of low density lipoprotein cholesterol (LDL), initiated in healthy young to middle aged adults can eliminate or markedly reduce the composite endpoint of incident all cause mortality, myocardial infarction, stroke or coronary revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Men 35-50 years of age
* Women 45 - 59 years of age (must be sterile or >2 years postmenopausal)
* LDL cholesterol greater than 1.8 mmol/L (70 mg/dL) based on testing performed within 1 year
* One risk factor for Coronary Heart Disease other than lipid abnormality:
* Obesity and hypertension [BP >140 mmHg systolic and waist circumference > 100 cm in men and >90 cm in women]
* family history of premature myocardial infarction [<60 years]
* South Asian ethnic history
* currently smoking

Exclusion Criteria:

* Currently taking cholesterol lowering medication
* Qualify for cholesterol lowering medication based on current guidelines
* Significant renal dysfunction (creatinine clearance <30 ml/min)
* Significant hepatic dysfunction (AST/ALT >2.0 times upper limit of normal)
* Active malignancy
* Diabetes
* Progressive or terminal illness, or other condition in which subject is unlikely to survive the study period
* Known allergy, hypersensitivity (anaphylaxis) ar adverse reaction to any statin
* Participation in a clinical trial (except observational studies) within previous 30 days
* Received any investigation product within 30 days prior to participation in this clinical trial
* Previously enrolled in this clinical trial

Ages: 35 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Time to first occurrence of myocardial infarction, revascularization, stroke or death from any cause in the follow up period | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr Michael Farkouh, MD, FRCPC, MSc, FACC, Principal Investigator — Peter Munk Cardiac Centre, University Health Network; Michael J Domanski, MD, Principal Investigator — University of Maryland, Baltimore
Locations (3):
- Canada (3):
  - Dr. Killian De Blacam Family Medical Practice, Greater Sudbury, Ontario
  - Dr. Gregory Garrioch Family Medical Practice, Greater Sudbury, Ontario
  - Dr. Reena Dhatt, Greater Sudbury, Ontario

REFERENCES:
- [Derived] Domanski MJ, Fuster V, Diaz-Mitoma F, Grundy S, Lloyd-Jones D, Mamdani M, Roberts R, Thorpe K, Hall J, Udell JA, Farkouh ME. Next Steps in Primary Prevention of Coronary Heart Disease: Rationale for and Design of the ECAD Trial. J Am Coll Cardiol. 2015 Oct 20;66(16):1828-1836. doi: 10.1016/j.jacc.2015.08.857. PMID 26483108